CLINICAL TRIAL: NCT04944524
Title: Randomized Trial of Tofacitinib Versus Methotrexate for Maintenance Therapy in Granulomatosis With Polyangiitis
Brief Title: Comparison of Tofacitinib and Methotrexate in the Maintained Treatment of GPA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TofMTX-GPA maintain
Record Dates: First submitted 2021-06-22; First posted 2021-06-29 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Granulomatosis With Polyangiitis
MeSH Terms: conditions — Granulomatosis with Polyangiitis | interventions — tofacitinib; Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tofactitinib (Experimental): partcipants would be given one tablet of tofacitinib (5mg per tablet), twice per day, the treatment duration will last 12 months during the whole follow-up period.
  Interventions: Drug: Tofacitinib
- Methotrexate (Active Comparator): partcipants would be given tablets of methotrexate (2.5mg per tablet) from the initial dose of 15mg (6 tablets) and add to the maximal and optimal dose of 20mg (8 tablets), once per week, the treatment duration will last 12 months during the whole follow-up period.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Tofacitinib — 1. Tofacitinib 5mg twice a day for 12months;
  2. Basic treatment with prednisone. (1) the initial dose of prednisone (or equivalent): 0.8mg/kg/day. (2) Glucocorticoids tapering: after two weeks' usage of initial glucocorticoids dose, glucocorticoids can be tapered if there's no disease activity (BVAS/WG=0) or at least 50% reduction of BVAS/WG and no new manifestations. Prednisone (or equivalent) was reduced to 10mg/d at the time of randomization.
  Other Names: Tof
  Arms: Tofactitinib
Drug: Methotrexate — 1. Methotrexate (15 mg/week initially and progressively increased every week by 2.5 mg, to a maximum and optimal dose of 20 mg/week)
  2. Basic treatment with prednisone. (1) the initial dose of prednisone (or equivalent): 0.8mg/kg/day. (2) Glucocorticoids tapering: after two weeks' usage of initial glucocorticoids dose, glucocorticoids can be tapered if there's no disease activity (BVAS/WG=0) or at least 50% reduction of BVAS/WG and no new manifestations. Prednisone (or equivalent) was reduced to 10mg/d at the time of randomization.
  Other Names: MTX
  Arms: Methotrexate

SUMMARY:
The aim of this study is to identify the optimal maintenance therapy for granulomatosis with polyangiitis (GPA) by comparing the MTX (standard regimen) with Tofacitinib in terms of efficacy, i.e. in preventing relapses.

DETAILED DESCRIPTION:
Granulomatosis with polyangiitis (GPA), a systemic small-vessel vasculitis, could involve multiple tissues and organs. Remission of GPA can be obtained in approximately 80% of the patients with a combination of corticosteroids and cyclophosphamide. However, relapses are frequent and remain a challenge. The optimal drug for maintenance treatment is not determined. Tofacitinib is a Jak inhibitor which has been proved to be effective in multiple inflammatory diseases such as rheumatoid arthritis. But the efficiency and safety of tofacitinib in treating GPA remains unclear yet. In the present randomized trial, the comparison of MTX (standard regimen) with Tofacitinib in terms of efficacy, i.e. in preventing relapses will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed or relapsing Granulomatosis with polyangiitis met the criteria of 1990 ACR and 2012 Chapel Hill criteria
2. Patients in disease flare have achieved remission using a treatment combining corticosteroids and IV cyclophosphamide
3. Remission is defined as a Birmingham Vasculitis Activity/ Wegener's granulomatosis (BVAS/WG) score of 0 and receiving 10 mg/day of oral prednisone (or equivalent) at least 2 weeks
4. Age 18 to 75 years
5. Written informed consent obtained before taking part in the study

Exclusion Criteria:

1. Severe GPA defined as potentially organ- or life-threatening disease (i.e. alveolar haemorrhage, heart failure caused by myocarditis or pericarditis, progressive neurological symptoms, deaf, blindness, et al.)
2. Serum creatinine>120umol/L or proteinuria>1.0g/d
3. Failure to response after treatment with methotrexate or cyclophosphamide previously
4. Receipt of a JAKi therapy previously
5. Co-existence of another systemic autoimmune disease
6. Secondary vasculitis (following neoplastic disease, an infection or antithyroid drugs)
7. Malignancy or history of malignancy
8. Infection by HIV, HCV, HBV or tuberculosis
9. Severe uncontrolled cardiovascular, pulmonary, liver, gastrointestinal, endocrine, hematological, neurological, or psychiatric diseases that are not related to systemic vasculitis
10. Allergic to any of the medication (cyclophosphamide, corticosteroids, tofacitinib, methotrexate)
11. Blood dyscrasias including confirmed: Hemoglobin <9 g/dL or Hematocrit <30%; White blood cell count <3.0 x 109/L; Absolute neutrophil count <1.5 x 109/L; Platelet count <100 x 109/L; Alanine transaminase or aspartate aminotransferase or total bilirubin>1.5 upper normal limit; Estimated glomerular filtration rate<60ml/min/1.73m2
12. Any medical or psychiatric disorder which, in the investigator's opinion, may prevent the administration of treatment and patient follow-up according to the protocol, and/or which may expose the patient to a too greater risk of an adverse effect.
13. Incapacity or refusal to understand or sign the informed consent form.
14. Pregnancy, breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Relapse rate (major or minor) at 12 months | From the enrollment to the the end of 12 month.
  The major or minor relapse rate equals to the patients with relapse/ total participants ( A major relapse should be defined as the re-occurrence or new onset of potentially organ- or life-threatening disease activity that cannot be treated with an increase of GC alone and requires further escalation of treatment. All other relapses should be classified as minor.)

SECONDARY OUTCOMES:
Time to first relapse. | From the enrollment to the the end of 12 month.
  The time period from the baseline to the time when the first relapse occurred.
Number of relapse | From the enrollment to the the end of 12 month.
  Total times of relapse during the whole period of 12-month follow-up.
Cumulative dosage of corticosteroids | From the enrollment to the the end of 12 month.
  The cumulative dosage of corticosteroids during the whole period of 12-month follow-up. The cumulative dosage = Sum of different dose of prednisone every day.
Adverse events | From the enrollment to the the end of 12 month.
  All the kinds of adverse event related to the treatment and the disease itself will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lindi Jiang, PhD, Study Chair — Fudan University
Locations (1):
- Department of Rheumatology in Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No